CLINICAL TRIAL: NCT04873557
Title: Copper Use as Protection Against Antimicrobial Resistance in the ICU
Acronym: CUPRIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad del Desarrollo (Other)
Responsible Party: Principal Investigator, Jose M Munita, Principal Investigator, Universidad del Desarrollo
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: CUPRIC001
Record Dates: First submitted 2020-11-25; First posted 2021-05-05 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Healthcare Associated Infection
Keywords: Healthcare Associated Infection; Multidrug-Resistant Organism; Carbapenem-resistant Enterobacterial; Methicillin-resistant Staphylococcus aureus; Vancomycin-Resistant Enterococcus; Intensive Care Unit
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Copper Intervention (Experimental): Intervention with copper-based surfaces plus copper-enriched linen
  Interventions: Other: Copper-based surfaces plus copper-enriched linen
- Control Group (No Intervention): Control group without copper intervention

INTERVENTIONS:
Other: Copper-based surfaces plus copper-enriched linen — We will assess the efficacy of our intervention to decrease the acquisition of nasal and intestinal colonization with MDROs and the development of HAIs in the ICU setting.
  Arms: Copper Intervention

SUMMARY:
CUPRIC is an investigator initiated and conducted, prospective, quasi-experimental study to determine whether the combined use of copper-alloyed objects plus copper-enriched textiles reduce the burden of MDRO colonization and HAIs incidence in the critically ill population.

DETAILED DESCRIPTION:
BACKGROUND: Healthcare-associated infections (HAI) are among the leading causes of preventable death and are associated with significant financial costs. Treatment of HAI has been complicated by the rise of antimicrobial resistance (AMR). AMR limits the number of effective antibiotics available to treat HAI. Therefore, the prevention of these infections is increasingly important. Current evidence indicates that patients' colonization with multidrug-resistant organisms (MDRO) is a critical issue with the potential of causing serious harm. Fortunately, newer strategies such as copper usage in the healthcare environment are under development and these approaches may decrease the burden of MDRO without disrupting gastrointestinal colonization resistance. This project will explore a cutting-edge strategy to decrease HAIs through the reduction of environmental reservoirs by replacement of high-touch surfaces and textiles in an intensive care unit (ICU) setting using the inherent antimicrobial properties of copper alloys. By studying the incidence of MDRO colonization of patients and rates of HAIs in patients exposed and unexposed to copper-based surfaces and textiles, the aim is to expand knowledge, to help optimize the practice of the application of antimicrobial surfaces in the ICU setting.

AIM: To establish the efficacy of the combined use of copper alloy-surfaced objects and copper-enriched textiles to reduce the burden of patients' MDRO colonization in the ICU.

METHODS: The investigators will conduct a prospective, quasi-experimental study in the ICU at the Hospital Regional de Iquique. During the first stage of the study (6 months), the investigators will determine the cumulative incidence of MDRO acquisition (primary outcome) and the incidence rate of HAIs in patients admitted to the ICU before installation of the antimicrobial copper products. During the second stage (6 months), the investigator will assess study outcomes after the installation of copper surfaces over highly touched surfaces within the patient unit.

EXPECTED RESULTS: It is expected a 30% reduction of the cumulative incidence of MDRO acquisition with respect to the control group. The investigators also expect this reduction to translate into a decrease of HAIs in the treatment versus the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age ≥18 years)
2. ≥ 72 h in the ICU
3. Provide informed consent (or via an appropriate proxy, according to local requirements).

Exclusion Criteria:

(a) Patients with conditions that preclude rectal or nasal sampling, such as total colectomy with a colostomy bag, facial surgery/trauma with nasal involvement, among others.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
MDRO acquisition | 12 months
  To determine the cumulative incidence of MDRO acquisition in patients admitted to the ICU before and after installation of antimicrobial copper surfaces and copper-enriched textiles.

SECONDARY OUTCOMES:
Incidence Rate of HAIs | 12 months
  To determine the incidence rate of HAIs in patients admitted to the ICU before and after installation of antimicrobial copper surfaces and copper-enriched textiles.
Incidence of acquisition of individual bacterial organisms | 12 months
  To determine the cumulative incidence of acquisition of individual bacterial organisms of interest before and after installation of antimicrobial copper surfaces and copper-enriched textiles.
Individual HAI development | 12 months
  To determine the cumulative incidence of development of each of the included HAIs separately (See 3.2.1), before and after installation of antimicrobial copper surfaces and copper-enriched textiles.

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Munita, MD, Principal Investigator — Universidad del Desarrollo
Locations (1):
- Hospital Regional de Iquique, Iquique, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haque M, Sartelli M, McKimm J, Abu Bakar M. Health care-associated infections - an overview. Infect Drug Resist. 2018 Nov 15;11:2321-2333. doi: 10.2147/IDR.S177247. eCollection 2018. PMID 30532565
- [Background] Salgado CD, Sepkowitz KA, John JF, Cantey JR, Attaway HH, Freeman KD, Sharpe PA, Michels HT, Schmidt MG. Copper surfaces reduce the rate of healthcare-acquired infections in the intensive care unit. Infect Control Hosp Epidemiol. 2013 May;34(5):479-86. doi: 10.1086/670207. PMID 23571364
- [Background] Schmidt MG, von Dessauer B, Benavente C, Benadof D, Cifuentes P, Elgueta A, Duran C, Navarrete MS. Copper surfaces are associated with significantly lower concentrations of bacteria on selected surfaces within a pediatric intensive care unit. Am J Infect Control. 2016 Feb;44(2):203-9. doi: 10.1016/j.ajic.2015.09.008. Epub 2015 Nov 6. PMID 26553403
- [Background] Tamma PD, Kazmi A, Bergman Y, Goodman KE, Ekunseitan E, Amoah J, Simner PJ. The Likelihood of Developing a Carbapenem-Resistant Enterobacteriaceae Infection during a Hospital Stay. Antimicrob Agents Chemother. 2019 Jul 25;63(8):e00757-19. doi: 10.1128/AAC.00757-19. Print 2019 Aug. PMID 31138574
- [Background] Kourbatova EV, Halvosa JS, King MD, Ray SM, White N, Blumberg HM. Emergence of community-associated methicillin-resistant Staphylococcus aureus USA 300 clone as a cause of health care-associated infections among patients with prosthetic joint infections. Am J Infect Control. 2005 Sep;33(7):385-91. doi: 10.1016/j.ajic.2005.06.006. PMID 16153484
- [Background] Sickbert-Bennett EE, DiBiase LM, Willis TM, Wolak ES, Weber DJ, Rutala WA. Reduction of Healthcare-Associated Infections by Exceeding High Compliance with Hand Hygiene Practices. Emerg Infect Dis. 2016 Sep;22(9):1628-30. doi: 10.3201/eid2209.151440. PMID 27532259
- [Background] Karpanen TJ, Casey AL, Lambert PA, Cookson BD, Nightingale P, Miruszenko L, Elliott TS. The antimicrobial efficacy of copper alloy furnishing in the clinical environment: a crossover study. Infect Control Hosp Epidemiol. 2012 Jan;33(1):3-9. doi: 10.1086/663644. Epub 2011 Dec 7. PMID 22173515
- [Background] Madden GR, Heon BE, Sifri CD. Effect of copper-impregnated linens on multidrug-resistant organism acquisition and Clostridium difficile infection at a long-term acute-care hospital. Infect Control Hosp Epidemiol. 2018 Nov;39(11):1384-1386. doi: 10.1017/ice.2018.196. Epub 2018 Sep 20. PMID 30231949
- [Background] Schmidt MG, Attaway HH, Sharpe PA, John J Jr, Sepkowitz KA, Morgan A, Fairey SE, Singh S, Steed LL, Cantey JR, Freeman KD, Michels HT, Salgado CD. Sustained reduction of microbial burden on common hospital surfaces through introduction of copper. J Clin Microbiol. 2012 Jul;50(7):2217-23. doi: 10.1128/JCM.01032-12. Epub 2012 May 2. PMID 22553242